CLINICAL TRIAL: NCT03040375
Title: Integrating Infant Feeding Counselling With Psychosocial Stimulation
Brief Title: Integrating Infant Feeding Counselling With Psychosocial Stimulation to Improve Child Growth and Development in Urban Slum of Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PR-14091
Record Dates: First submitted 2016-12-27; First posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2014-11

CONDITIONS: Infant Malnutrition; Cognitive Change
MeSH Terms: conditions — Infant Nutrition Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peer counselling (Experimental): There were two types of intervention: one providing breast-feeding and complementary feeding counselling + psychosocial stimulation interventions.
  Interventions: Behavioral: Peer counselling
- Non peer counselling (No Intervention): Usual health messages

INTERVENTIONS:
Behavioral: Peer counselling
  Arms: Peer counselling

SUMMARY:
Undernutrition and poor cognitive development affect many children under 5 in developing countries, who are exposed to multiple risk factors including poverty, malnutrition, poor health, and unstimulating home environments. The optimum development and growth of young children requires affection and responsiveness from the mother/caregiver, cognitive stimulation, good nutrition and infection control. In Bangladesh, stimulation at home is generally poor and contributes to children's poorer development. It is important to show that psychosocial stimulation programmes through home visits integrated into the feeding programmes can benefit children's growth and development. This study will help to fill this evidence gap about effective interventions to improve infant and young child growth and development in Bangladesh. Considering the high prevalence of undernutrition and low prevalence of stimulating environments in Bangladesh, it is important to show evidence that integrating infant feeding counselling and psychosocial stimulation activities result in optimum child growth & development. To determine if combined infant feeding counselling and psychosocial stimulation programme (promoting mothers positive parenting) starting in the 3rd trimester of pregnancy, further improves: children's cognitive, motor and language development along with growth and mothers' child rearing and child-feeding knowledge and practices compared to peer counselling alone or usual health messages only. We used a community-based CRCT to examine the impact of a peer counselling infant feeding education program with psychosocial stimulation starting in the third trimester of pregnancy to one year after delivery, to improve child growth and cognition, language, behaviour and psychomotor development compared to a control group receiving usual health messages. The outcome assessments were made on a cohort of infant-mother dyads measured at baseline and at follow up visits. Outcome assessments were conducted with all the mother-infant pairs recruited in the community clusters in the study, with an expected total of 334 mother-infant dyads (167 in each treatment group).The main outcomes are children's growth, cognition, language, behaviour and psychomotor development

DETAILED DESCRIPTION:
Study design It was a randomized controlled trial of integrating infant feeding counselling and psychosocial stimulation in slums of Mirpur, Dhaka. The trial was conducted in slum communities on the edge of Dhaka with 10 clusters of city blocks for each of the 2 study groups (167 mothers/infant pairs in each group). The two groups 1) Psychosocial stimulation + feeding counselling group and 2) Control group. The peer counselling education and psychosocial stimulation intervention will be delivered to the mothers, by locally recruited and trained peer counsellors, starting in the third trimester of pregnancy until the child is one year of age. The peer counselling education was offered to eligible pregnant women identified by household survey over 2 months in each community cluster in the intervention groups. Using a similar approach to recruitment, a cohort of mother-infant dyads, who received standard maternal and child health care programmes,were identified in the control clusters. Outcome assessments conducted with all the mother-infant pairs recruited in the community clusters in the study, with an expected total of 334 mother-infant dyads. There was a baseline assessment of demographic information and further assessments of growth every 3 months from birth until the children are 12 months of age. The developmental assessments in children will be conducted at 12 months of age.

Sampling scheme A community based randomized controlled trial namely "Mirpur Shishu Pushti Trial" is ongoing in 36 clusters within 4 wards of Mirpur municipality. The average population of a "Ward" is 350,000 people. There are approximately five "Mahallas" per "Ward" with an average population of 70,000 people. The unit of randomization for this trial was city block clusters (CBC) with a population of about 6,000. A list of 36 CBC has already been prepared using established GIS methods to map and census the households. These CBC are being used in the ongoing community trial (Shishu Pusti trial). This ongoing study includes two arms; a peer-counselling (Infant and Young Child Feeding) arm and a control arm and the aims are to assess if the peer-counselling program improves children's growth through an improvement in child-feeding program. In this present study, two stage cluster sampling will be used, at the first stage 10 cluster will be randomly selected from 36 pre-defined clusters under this study area, on the second stage, 5 clusters will be randomly allocated for each of the treatment group. As the duration of the present study is only 18 months, utilization of the same study field along with GIS mapping and population census will allow us to minimize time as well as cost for the current study.

Trained field assistants identified women who were in their third trimester of pregnancy by systematic door-to-door surveys across the "clusters" over two months period. Pregnant women aged 16 to 49 years were included. Women who plan to migrate from the Mirpur area after delivery was excluded.

There will be two types of intervention: one providing breast-feeding and complementary feeding counselling and the other breast-feeding and complementary feeding counselling + psychosocial stimulation interventions. The proposed individual peer counselling education will be of sufficient intensity to alter infant and young child feeding practices and to improve the growth and development of the young children, hence prevent malnutrition and developmental delay. The interventions will be delivered to the women starting in last trimester of pregnancy and until their child is one year of age.

a. Description of intervention

The approach to promoting appropriate infant and young child feeding was through a programme of home-based peer counselling by trained, local women from the mothers' community. The peer counselling education and psychosocial stimulation intervention delivered to the mothers, by Peer Counsellors. The stimulation intervention included age-appropriate developmental messages and handmade toys provided by the Counsellors during home visits at regular intervals along with feeding counselling. The mothers were shown age appropriate stimulation activities for their child. There was at least 13 visits by the Counsellors: 2 visits before delivery; 2 visits during the 1st month; 7 monthly visits between age 2 to 8 months; and 2 visits at age 10 and 12 months and bi-weekly group meetings. The integrated programme included social mobilization activities to help families adapt improved child care practices to achieve optimum child growth and development.

i) Selection and training of peer counsellors Women with personal breastfeeding experience, at least 6 years of schooling, residing in the same area, and motivated to work were selected to become peer counsellors. The WHO/UNICEF Breastfeeding Counselling Course adapted to the local language and culture, which has already been validated in a previous study, was used for training of peer counsellors. The training was given for 40-h (4-h daily for 10 days). Counselling skills was taught mainly by demonstrations and role play and included: listening to mothers, learning about their difficulties, assessing the position and attachment of babies during breastfeeding, building mother's confidence, giving support and providing relevant information and practical help when required. During the training course antenatal and postpartum counselling wase practiced with pregnant women, mothers with newborns and infants aged 1-12 months in the field site. The counsellors were also be taught how to use locally available foods for complementary feeding of infants and young children, and how best to demonstrate these food preparation skills to mothers.

The stimulation intervention included age-appropriate developmental messages, flip charts and handmade toys that will be provided by the Peer Counsellors during home visited at regular intervals along with feeding counselling. The mothers were shown three to four age appropriate stimulation activities with child and how to make toys using recycled materials. As children grow up, mothers were also be taught how to make simple one page books, suitable for use by less literate mothers.

The short version of the Stimulation Curriculum will take 30-40 minutes and included the following activities during home visits

* Explaining 2-3 stimulation messages (e.g. how to show love, how to respond, how to facilitate communication etc) along with their benefits on child-development
* Explaining 1 Pictorial Stimulation Calendar containing 3 to 4 age appropriate activities with the child until next visit
* Teaching mothers and other family members how to make toys from recycled materials The performance of the counsellors was monitored at least four times during the course of the study by the Senior Infant Feeding Counsellors and stimulation supervisors.

ii) Counseling schedules: There was a schedule of at least 13 visits by the peer counsellors: two before delivery; two during the first month; seven monthly visits between age 2 to 8 months; and two visits at age 10 and 12 months. The counselling took place at home to ensure key family members (e.g. mother-in-law and fathers) can also be included in the counselling sessions. The duration of each visit was from 30 to 40 minutes.

Antenatal visits: The peer counsellors during the two antenatal contactswould prepare the mothers, and other members of the family who would support her at delivery, about the importance of holding the baby within a few minutes of delivery and how to initiate breastfeeding within one hour of delivery.

In addition, they would provide some guidelines on the importance of feeling well and happy during pregnancy, singing to the baby in the womb, avoiding any harmful practices like use of tobacco. Fathers and other household members was be briefed on the importance of keeping the mother happy and joyful and avoiding subjecting her to violence or any harsh treatment. ECD messages like playing, chatting and singing to the newborn will be provided in the psychosocial stimulation arm along with feeding messages.

Visits in the first month of life: The mothers were contacted twice by the peer counsellors (within 48 hours of delivery and at 10-14 days). At these visits exclusive breastfeeding was encouraged and the mother's specific needs addressed. Issues that could be covered include sore nipples, problems with attachment to the breast, the baby's position during feeds, family pressure to start other foods and mothers' doubts about the adequacy of their breast milk. I Age-appropriate ECD messages was provided and mothers will be prepared for child's developmental requirements as s/he grows.

Visits 2 to 8 months of life: The mothers were contacted monthly by the peer counsellors. Specific problems will be addressed and continued support for breastfeeding provided especially how to deal with pressures to introduce other foods and concerns about the adequacy of the growth of the infant. From 6 months of age, specific messages that include, the importance of complementary feeding, demonstration and preparation of complementary foods introduction. Mothers will be given measuring cups and spoons and appropriate complementary foods were demonstrated and use of usual foods in the home will be encouraged.

Similarly other age-appropriate ECD messages was provided and PCs will try to include other family members in these sessions.

Visits at 10 and 12 months of life: The mothers contacted at 10 and 12 months by the peer counsellors. The mothers were encouraged to continue breastfeeding and support will be given for adequate frequency of complementary feeds and appropriate diversity foods.

ELIGIBILITY:
Inclusion Criteria:

* women aged 16 to 49 at third trimester pregnancy
* No medical record of chronic disease
* who would stay next 1 year in the study area
* Healthy neonate

Exclusion Criteria:

* Women having reported chronic illness
* Would not stay in the study area
* extremely low birth weight neonate
* neonate with congenital anomaly

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2014-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Changes in percentage of motor development among the children at 9 &12 months who received intervention | 9 and 12 months
Early Initiation of Breastfeeding rate | from birth to every 2 months till 1 year
Differences in percentage of stunting, wasting and underweight among the children who received intervention | from birth to every 2 months till 1 year

SECONDARY OUTCOMES:
Differences in percentage of children at 6 & 9 months who receive solid, semi-solid or soft foods. | 6 to 12 months
Differences in percentage of children consuming foods from >4 food groups | 6 to 12 months
Differences in the mean intake of food energy, protein, carbohydrate, fat and selected micronutrients from complementary feeds | 6 to 12 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ara G, Khanam M, Papri N, Nahar B, Kabir I, Sanin KI, Khan SS, Sarker MSA, Dibley MJ. Peer Counseling Promotes Appropriate Infant Feeding Practices and Improves Infant Growth and Development in an Urban Slum in Bangladesh: A Community-Based Cluster Randomized Controlled Trial. Curr Dev Nutr. 2019 Jun 18;3(7):nzz072. doi: 10.1093/cdn/nzz072. eCollection 2019 Jul. PMID 31334480